CLINICAL TRIAL: NCT06645600
Title: Are Balance and Lower Extremity Muscle Strength Indicators of Fracture Risk Independently of Bone Mineral Density in Postmenopausal Women?: a Cross-sectional Study
Brief Title: Balance and Muscle Strength as Indicators of Fracture Risk in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principal Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikdüzüStateH3
Record Dates: First submitted 2024-09-28; First posted 2024-10-17 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fracture risk — To calculate fracture risk, the percentages for major and hip fracture risks will be calculated using the Fracture Risk Assessment Tool (FRAX®). The one-leg stance test, used to assess static posture and balance, and the 30-second sit-to-stand test, used to evaluate endurance and lower extremity strength, will be applied to the patients.

SUMMARY:
The study is designed as a cross-sectional clinical study. A total of 156 postmenopausal women who visited the Physical Therapy and Rehabilitation outpatient clinic at Beylikdüzü State Hospital and have had Dual X-ray Absorptiometry (DXA) measurements taken within the last 6 months will be included. The sociodemographic data of the patients will be recorded. Femoral neck and lumbar L1-L4 T-scores and femoral neck bone mineral density (BMD) values obtained from DXA measurements will be collected. To calculate fracture risk, the percentages for major and hip fracture risks will be calculated using the Fracture Risk Assessment Tool (FRAX®). The one-leg stance test, used to assess static posture and balance, and the 30-second sit-to-stand test, used to evaluate endurance and lower extremity strength, will be applied to the patients.

DETAILED DESCRIPTION:
This study is designed as a cross-sectional clinical investigation aimed at assessing fracture risk in postmenopausal women. A total of 156 postmenopausal women who attended the Physical Therapy and Rehabilitation outpatient clinic at Beylikdüzü State Hospital and had undergone Dual X-ray Absorptiometry (DXA) measurements within the past six months will be included. Sociodemographic data, such as age, weight, height, and medical history, will be recorded for each participant.

The study will gather femoral neck and lumbar L1-L4 T-scores, as well as femoral neck bone mineral density (BMD) values, obtained from DXA scans. To evaluate the risk of fractures, major and hip fracture percentages will be calculated using the Fracture Risk Assessment Tool (FRAX®), a widely accepted method for predicting fracture risk in osteoporosis patients.

Two functional tests will be applied: the one-leg stance test, which measures static balance and postural stability, and the 30-second sit-to-stand test, which assesses lower extremity strength and endurance. These simple, quick tests will be used to determine whether they can serve as practical predictors of fracture risk in postmenopausal patients. The study aims to evaluate whether these two functional tests can provide rapid and effective fracture risk assessments in clinical practice, offering a valuable tool for clinicians in identifying high-risk patients early and implementing preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* Being a postmenopausal woman over the age of 50,
* Agreeing to participate in the study,
* Having no conditions that would prevent the individual from performing the tests to be administered during the study.

Exclusion Criteria:

* Refusal to participate,
* Presence of neuromuscular or cardiac diseases that would prevent the performance of the tests,
* Psychiatric disorders,
* Cognitive impairments,
* Uncontrolled hypertension,
* Use of medications that could affect the study results.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: postmenopausal women
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
The one-leg stance test score | 0 day
  The one-leg stance test is a simple and widely used balance assessment tool. During the test, the individual is asked to stand on one leg while maintaining balance for as long as possible without support. The test is typically performed with eyes open, and the duration for which the person can remain stable on one leg is recorded. It helps evaluate static balance and postural control, and poor performance on the test can be indicative of an increased risk of falls or fractures, particularly in older adults or those with musculoskeletal issues.
The 30-second sit-to-stand test score | 0 day
  The 30-second sit-to-stand test is a functional assessment tool used to evaluate lower extremity muscle strength and endurance. During the test, the individual is asked to sit in a standard chair and then stand up and sit down as many times as possible within 30 seconds. The number of complete stands is recorded. This test is commonly used to assess functional mobility and leg strength, particularly in older adults or those with conditions affecting muscle function. It provides a quick and practical measure of lower body strength, which is important for daily activities and fall prevention.

SECONDARY OUTCOMES:
FRAX Hip and Major Fracture Risc | 0 day
  FRAX (Fracture Risk Assessment Tool) is a widely used algorithm developed by the World Health Organization (WHO) to estimate an individual's 10-year probability of experiencing a major osteoporotic fracture (hip, spine, forearm, or shoulder) and hip fracture specifically. It is designed to help clinicians assess fracture risk in patients, especially those with osteoporosis or low bone mineral density (BMD), and guide decisions regarding the need for interventions like pharmacological treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Şirin Ahısha, MD, Principal Investigator — Beylikdüzü State Hospital
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Beylikdüzü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No